CLINICAL TRIAL: NCT04890951
Title: Prospective Multi-site Cohort Study Investigating Hysterectomy Versus Uterine Preservation for Pelvic Organ Prolapse Surgery: The HUPPS Study
Brief Title: Hysterectomy Versus Uterine Preservation for Pelvic Organ Prolapse Surgery
Acronym: HUPPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The MSI Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: REB19-2134
Record Dates: First submitted 2021-05-05; First posted 2021-05-18 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic Organ Prolapse; Gynecologic Surgery; Female; Epidemiology
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Hysterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uterine Preservation
  Interventions: Procedure: Hysteropexy
- Hysterectomy
  Interventions: Procedure: Hysterectomy and vaginal vault suspension

INTERVENTIONS:
Procedure: Hysteropexy — Uterine preservation through suspension
  Groups: Uterine Preservation
Procedure: Hysterectomy and vaginal vault suspension — Uterine removal and sewing the vagina upwards
  Groups: Hysterectomy

SUMMARY:
Pelvic organ prolapse (POP) is the descent of pelvic organs into the vagina resulting in bulge symptoms and occurs in approximately 50% of women. Almost 20% of women will elect surgical correction of this condition by age 85. Removal of the uterus (hysterectomy) with concomitant vaginal vault suspension is a longstanding practice in POP surgery to address apical (uterine) prolapse. Yet, contemporary evidence on the merits of this approach relative to preservation of the uterus through suspension is needed to better inform surgical decision-making by patients and their healthcare providers. The objective of this trial is to evaluate POP-specific health outcomes and service utilization of women electing uterine suspension compared to those electing hysterectomy and vaginal vault suspension for POP surgery up to 1-year post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Have diagnosed POP of stage ≥2 using the globally recognized Pelvic Organ Prolapse-Quantification System (POP-Q)
* Elect surgical management of POP
* Demonstrate presence of apical prolapse on clinical exam deemed to require either a hysterectomy and concomitant vaginal vault suspension or uterine suspension to properly address their POP during surgical correction
* Desire no further pregnancy
* Can communicate in English
* Are ≥18 years in age

Exclusion Criteria:

* Prior hysterectomy

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women seeking surgical correction of POP at one of the study sites.
Sampling Method: Probability Sample
Enrollment: 321 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Anatomic failure to correct apical POP | 1 year
  Descent of the apex (POP-Q point C) equal to or beyond one half of the total vaginal length

SECONDARY OUTCOMES:
Overall failure to correct POP | 1 year
  POP-Q stage ≥2 in any compartment, or re-treatment of POP with physiotherapy, pessary, or repeat surgery
Subjective failure to correct POP | 6 weeks; 1 year
  Patient report of bulge symptoms at 6 weeks or 1 year, using one item on the PFDI-20: "Do you usually have a bulge or something falling out that you can see or feel in the vaginal area?"
Length of surgery (minutes) | Peri-operative
Estimated blood loss during surgery >500 mL | Peri-operative
Procedural complications | Peri-operative
  E.g., peri-operative blood transfusion, visceral injury
Post-operative infection | Peri-operative
  E.g., abscess, urinary tract infection
Opioid use in-hospital | Peri-operative
  Measured by Morphine milliequivalent (mEq)
Resumption of spontaneous voiding (days) | Peri-operative
Length of post-operative stay (days) | Peri-operative
PROM: Total Pelvic Floor Impact Questionnaire-7 (PFIQ-7) score | 6 weeks; 1 year
  Change from baseline
PROM: Total POP Incontinence Sexual Questionnaire Revised (PISQ-IR) score | 6 weeks; 1 year
  Change from baseline
PROM: Total Pelvic Floor Distress Inventory-20 (PFDI-20) score | 6 weeks; 1 year
  Change from baseline
Presentation at the emergency department | 30 days (any health complaint); 1 year (pelvic floor-related complaint)
Hospital readmission | 30 days (any health complaint); 1 year (pelvic floor-related complaint)

CONTACTS AND LOCATIONS:
Locations (1):
- Pelvic Floor Clinic, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scime NV, Ramage K, Brennand EA; Calgary Women's Pelvic Health Research Group. Protocol for a prospective multisite cohort study investigating hysterectomy versus uterine preservation for pelvic organ prolapse surgery: the HUPPS study. BMJ Open. 2021 Oct 4;11(10):e053679. doi: 10.1136/bmjopen-2021-053679. PMID 34607873